CLINICAL TRIAL: NCT02896699
Title: Advanced HIV Prevention (PrEP Chicago)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB15-1250
Record Dates: First submitted 2016-07-26; First posted 2016-09-12 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: HIV
Keywords: Pre-exposure prophylaxis (PrEP); diffusion of innovation; men who have sex with men; LGBT; African American; Black; HIV; network analysis; network intervention
MeSH Terms: conditions — Homosexuality | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PrEP Intervention Group (Experimental): Group training session including HIV Education, PrEP Education, Following the training session Booster phone calls HIv and syphillis testing
  Interventions: Behavioral: PrEP Intervention Group
- Control Group (Active Comparator): Group HIV risk vignettes
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: PrEP Intervention Group
  Arms: PrEP Intervention Group
Other: Control Group
  Arms: Control Group

SUMMARY:
This study will evaluate the feasibility of a network intervention to train individuals to disseminate PrEP information and motivate initial PrEP interest and knowledge of PrEP in their social networks.

DETAILED DESCRIPTION:
The specific aims of this study are:

1. To recruit 450 participants in Chicago, Illinois, and to train them as peer change agents (randomized to cross-over groups) to disseminate PrEP information and motivate PrEP interest and knowledge of PrEP in their local networks.
2. To evaluate feasibility of the program over 2 years of participant follow-up through: 1) peer change agent exit survey; 2) peer change agent booster sessions; 3) peer change agent communication with University of Chicago PrEP program social media; 4) referrals into the project and; 5) calls into the PrEP warmline.

ELIGIBILITY:
Inclusion Criteria:

* Lives on the South Side of Chicago, Illinois
* Born male
* Has had sex with men in the previous year
* Is an active Facebook user
* Does not have plans to leave Chicago

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 424 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Network member call into the PrEPline | 2 years

SECONDARY OUTCOMES:
PrEP Attitudes questionnaire | 2 years
  Monitor the change in attitude towards PrEP (1) from baseline measure to 12-months; (2) 12-months to 24-months; and (3) baseline to 24-month.
Peer change agent boosters sessions completed | 2 years
Number of Facebook posts with respect to PrEP and sexual health | 2 years
Number of referrals enrolled into the study | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young LE, Schumm P, Alon L, Bouris A, Ferreira M, Hill B, Khanna AS, Valente TW, Schneider JA. PrEP Chicago: A randomized controlled peer change agent intervention to promote the adoption of pre-exposure prophylaxis for HIV prevention among young Black men who have sex with men. Clin Trials. 2018 Feb;15(1):44-52. doi: 10.1177/1740774517730012. Epub 2017 Sep 1. PMID 28862483